CLINICAL TRIAL: NCT05332808
Title: Treatment State and Quality of Life in HIV- Infected Patients in Upper Egypt
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Saleem Zayan, MD, Assiut University
Other Study IDs: HIV patients characteristics
Record Dates: First submitted 2022-04-12; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnare — collecting data about treatment and quality of life

SUMMARY:
HIV stands for Human Immunodeficiency Virus, a pathogen that works by attacking the human immune system. It belongs to a class of viruses called retroviruses and more specifically, a subgroup called lentiviruses, or viruses that cause disease slowly.

In 2020, there were about 37.7 million people living with HIV. Only 84% of all people living with HIV knew their HIV status in 2020, with 680 000 people died from AIDS-related illnesses in 2020 .

HIV cannot replicate on its own, so in order to make new copies of itself, it must infect cells of the human immune system, called CD4 cells. . CD4 cells are white blood cells that play a central role in responding to infections in the body. Over time, CD4 cells are killed by HIV and the body's ability to recognise and fight some types of infection begins to decline If HIV is not controlled by treatment, the loss of CD4 cells leads to the development of serious illnesses, or 'opportunistic infections'. In people with normal CD4 cell levels, these infections would be recognised and cleared by the immune system.

Experiencing a collection of these infections is the most advanced stage of HIV, which is when a person is also said to have AIDS (Acquired Immune Deficiency Syndrome). Effective testing and treatment of HIV means that the large majority of people living with HIV do not reach this stage.

Stages of HIV :

An initial acute infection; (ii) a long asymptomatic period; and (iii) a final increase in viral load with a simultaneous collapse in healthy CD4+ T cell count during which AIDS appears During the acute infection period (2-10 weeks) there is a sharp drop in the concentration of circulating CD4+ T cells, and a large spike in the level of circulating free virus. Clinically the patient suffers from infectious mononucleosis-like systemic illness with fever, diarrhoea, often a transient meningo-encephalitis and even lung pneumocystosis .After this period, the level of circulating CD4+ T cells returns to ''near-normal'' levels, and the viral load drops dramatically. In this asymptomatic or latent period, the patient does not exhibit any major symptoms of disease, even though HIV is continuously infecting new cells and actively replicating. Normally this latent period ranges in duration from 7 to 10 years, Following this asymptomatic period, the viral load rises rapidly with a simultaneous drop in CD4+ T cell count. This last stage is called AIDS, and is defined by situations where CD4+ T cell counts are below 200 cells/mm3 or when certain opportunistic infections are experience Treatment for HIV Antiretroviral medicines are used to treat HIV. They work by stopping the virus replicating in the body, allowing the immune system to repair itself and preventing further damage. These come in the form of tablets, which need to be taken every day.

HIV is able to develop resistance to a single HIV medicine very easily, but taking a combination of different medicines makes this much less likely. Most people with HIV take a combination of medicines. It's vital these are taken every day as recommended by your doctor. The goal of HIV treatment is to have an undetectable viral load. This means the level of HIV virus in your body is low enough to not be detected by a test.

Quality of life of HIV infected patients:

Quality of life has been considered synonymous with health status, functional status, psychological wellbeing, happiness with life, satisfaction of needs, and assessment of one's own life . Assessment of quality of life has become an important outcome measure in the management of HIV/AIDS and reflects improvement or otherwise of the health experience and satisfaction with care among patients living with HIV/AIDS

ELIGIBILITY:
Inclusion Criteria:

* any HIV patient

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV patients at upper Egypt hospitals
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
completion of questionnaire | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Shimaa, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided